CLINICAL TRIAL: NCT05893381
Title: A Phase II Randomized Trial of Lu-PSMA and Stereotactic Radiotherapy Versus Radiotherapy Alone for Oligometastatic Prostate Cancer (LUST)
Brief Title: Lu-PSMA and Stereotactic Radiotherapy Versus Radiotherapy Alone for Prostate Cancer (LUST)
Acronym: LUST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST185.09
Record Dates: First submitted 2023-05-30; First posted 2023-06-07 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
Keywords: PSMA PET/CT positive
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic Radiotherapy followed by Lu-PSMA (arm A) (Experimental): Ablative stereotactic radiation on the metastatic sites. Delivered in a 1 to 5 fractions regimen. 177Lu-PSMA-I&T in 2 cycles of treatment at 6-8 weekly intervals at a dosage of 7.4 Gigabequerel (GBq)
  Interventions: Drug: [177Lu]Lu-PSMA I&T; Radiation: Stereotactic Radiotherapy
- Stereotactic Radiotherapy (arm B) (Active Comparator): Ablative stereotactic radiation on the metastatic sites. Delivered in a 1 to 5 fractions regimen.
  Interventions: Radiation: Stereotactic Radiotherapy

INTERVENTIONS:
Drug: [177Lu]Lu-PSMA I&T — The radiopharmaceutical 177Lu-PSMA-I&T will be administered, by slow intravenous injection, in 2 cycles of treatment at 6-8 weekly intervals at a dosage of 7.4 GBq.
  Other Names: 177Lu-PSMA
  Arms: Stereotactic Radiotherapy followed by Lu-PSMA (arm A)
Radiation: Stereotactic Radiotherapy — Ablative stereotactic radiation on the metastatic sites. Delivered in a 1 to 5 fractions regimen, depending on the target size and the surrounding normal tissue constraints,
  Other Names: Ablative stereotactic radiation

SUMMARY:
Multicenter, open-label, parallel-group, phase II randomized study in patients with oligometastatic prostate cancer with 1-3 asymptomatic metastases of the soft tissue or bone. Eligible patients will be randomized at 1:1 ratio to Stereotactic Radiotherapy followed by Lu-PSMA (arm A) or Stereotactic Radiotherapy (arm B)

DETAILED DESCRIPTION:
Biochemical recurrence (BCR), i.e. prostate-specific antigen (PSA) only recurrence occurs in nearly one-third of patients, after primary definitive therapy for prostate cancer.

PSMA (prostate-specific membrane antigen) is an attractive target for diagnosis and therapy of metastasized prostate cancer (PCa) as its expression levels are directly correlated with androgen independence, metastases and progression.

Positron Emission Tomography/Computed Tomography (PET-CT) using PSMA is able to detect > 50% of relapses with PSA between 0.50 and 1 ng/mL and >75% with PSA between 1 and 2.

Oligometastatic prostate cancer include 1-3 asymptomatic metastatic lesion(s) of the soft tissue or bone. The treatment of oligometastatic disease depends on multiple factors including the site, the size, number and location of metastases, and the effectiveness of treatments.

Recent advances in radiation therapy allow to image and treat precisely target lesions within any anatomic region of the body. Stereotactic radiation therapy permit highly conformal and precisely targeted radiation administered in a dose intensive strategy. Local control in excess of 75% has been reported for metastatic prostate cancer with very low toxicity.

Lutetium 177-PSMA (177Lu-PSMA) is the most extensively investigated PSMA radioligand for radionuclide therapy in castration resistant prostate cancer (CRPC). Several retrospective studies and three phase II prospective studies demonstrated safety and impressive efficacy of 177Lu-PSMA in metastatic CRPC (mCRPC).The purpose of this study is to evaluate in a randomized phase II study the impact of Lu-PSMA added to stereotactic radiotherapy vs radiotherapy alone in PSMA detected- metastatic lesions of hormone-sensible prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with prostate cancer must have 1-3 asymptomatic metastatic lesions that are ≤ 5.0 cm or < 250 cm3 documented at CT/MRI or WBD-MRI.
2. PSMA-PET/CT positive scan matching with lesions documented on baseline CT/MRI or WBD-MRI.
3. Patients must have had their primary tumor treated with surgery and/or radiation and previous salvage radiation to the prostate bed or pelvis is allowed.
4. Patients will be admitted to the therapeutic phase only if diagnostic PET/CT PSMA SUV max is ≥ 3.
5. Histologic confirmation of malignancy (primary or metastatic tumor).
6. Prostate specific antigen (PSA) ≥ 0.2 ng/mL but ≤ 50 ng/mL and Testosterone ≥ 125 ng/dL.
7. PSA doubling time (PSADT) < 15 months. PSADT will be calculated using as many PSA values that are available from time of relapse (PSA > 0.2 ng/dL).
8. Patients unfit or refusing ADT.
9. Patients may have had prior systemic therapy and/or ADT associated with treatment of their primary prostate cancer. Patients may have had ADT associated with salvage radiation therapy.
10. Patients must be ≥ 18 years of age.
11. Patient understands the purpose of the study and the procedures required for it; the patient is willing to participate in the study and to sign a written informed consent document.
12. Patients must have an Eastern Cooperative Oncology Group performance status ≤ 2.
13. Patients should have a life expectancy of at least 6 months.
14. Patients must have normal organ and marrow function as defined as:

    * Leukocytes >2,000/μL;
    * Absolute neutrophil count >1,000/μL;
    * Platelets >75,000/μL;
    * total bilirubin within normal institutional limits (this will not apply to patients with confirmed Gilbert's syndrome);
    * AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional upper limit of normal;
    * Creatinine within normal institutional limits.
15. If the participant engages in sexual activity with a woman of childbearing potential, a condom must be used together with another highly effective method of contraception during the Treatment Period and for 6 months after the last dose of study intervention. The participant must agree not to donate sperm for the purpose of reproduction during the Treatment Phase and for a minimum of 6 months after receiving the last dose of study intervention.
16. Highly effective birth control methods are required beginning at the screening visit and continuing until 6 months following last treatment with study drug. Patients and female partner who is of childbearing potential must use 2 acceptable methods of birth control (1 of which must include a condom as a barrier method of contraception, see Appendix F) starting at screening and continuing throughout the study period and for 6 months after final study drug administration. Two acceptable methods of birth control thus include Condom (barrier method of contraception) and one of the following is required ( established use of oral, or injected or implanted hormonal method of contraception by the female partner; placement of an intrauterine device (IUD) or intrauterine system (IUS) by the female partner; additional barrier method like occlusive cap with spermicidal foam/gel/film/cream/suppository in the female partner; tubal ligation in the female partner; vasectomy or other procedure resulting in infertility (eg., bilateral orchiectomy), for more than 6 months.

16. Highly effective birth control methods are required beginning at the screening visit and continuing until 6 months following last treatment with study drug. Patients and female partner who is of childbearing potential must use 2 acceptable methods of birth control (1 of which must include a condom as a barrier method of contraception, starting at screening and continuing throughout the study period and for 6 months after final study drug administration.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

1. No more than 3 years of ADT is allowed, with the most recent ADT treatment having occurred more than 6 months prior to enrollment.
2. PSMA -PET/CT scan more than 3 months.
3. Spinal cord compression or impending spinal cord compression.
4. Suspected pulmonary and/or liver metastases.
5. Bone metastasis in a femoral bone.
6. Previous radiation therapy on the metastatic site.
7. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. A window of 3 days is permitted.
8. Participation in another clinical trial with any investigational agents within 30 days prior to study screening. A window of 3 days is permitted.
9. Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant.
10. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
11. History of allergic reactions attributed to compounds of similar chemical or biologic composition to 177-Lu-PSMA- I & T or other agents used in the study.
12. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
13. Unable to lie flat during or tolerable SABR.
14. Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 3 years (except for previously treated basal cell carcinoma);
15. Known HIV-positivity, whether or not symptomatic.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
12-month PSA (Prostate-Specific Antigen)-progression-free survival (PSA-PFS) | 12-months
  To determine the proportion of men with oligometastatic hormone sensitive prostate cancer who have PSA progressed after 12 months from randomization to Stereotactic Radiotherapy and Lu-PSMA versus Radiotherapy alone.

SECONDARY OUTCOMES:
12-month radiographic Progression-free survival (rPFS), Androgen Deprivation Therapy-Free survival (ADT-FS) and Total progression-free survival (PSA-PFS+rPFS) | 12-months
  To assess radiographic progression free survival (PFS) after 12 months, ADT free survival (ADT-FS) and Total progression-free survival (PSA-PFS+rPFS) of Lu-PSMA + Stereotactic Radiotherapy vs Stereotactic Radiotherapy defined as the time interval between the day of randomization and the day of disease progression.
Incidence of Treatment-Emergent Adverse Events [Toxicity] | 60 months
  To describe the toxicity of Lu-PSMA + Stereotactic Radiotherapy vs Stereotactic Radiotherapy for the population enrolled using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Overall survival (OS) | 60 months
  To assess overall survival (OS) defined as the time interval between the day of randomization and death or last contact.
Proportion of subjects with undetectable PSA (<0.2 ng/mL) | 60 months
  To assess proportion of subjects with undetectable PSA (<0.2 ng/mL) defined as a PSA level ≤0.20 ng/mL as measured during routine follow-up
Quality of life questionnaire (QLQ) | 60 months
  To assess quality of life in the Lu-PSMA+ Stereotactic Radiotherapy arm vs Stereotactic Radiotherapy only arm using the Functional Assessment of Cancer Therapy - Prostate (FACT-P version 4) questionnaire. The scale ranging from 0-4, where 0 is labeled 'Not at all', and 4 is labeled 'Very Much'.

CONTACTS AND LOCATIONS:
Overall Officials: Federica Matteucci, Principal Investigator — UO Medicina Nucleare, IRCCS IRST
Locations (2):
- Italy (2):
  - UO Medicina Nucleare, AUSL della Romagna, Cesena, FC
  - UO Medicina Nucleare, IRCCS IRST, Meldola, FC